CLINICAL TRIAL: NCT04776902
Title: Effects of Ovarian Reserve on Sexual Satisfaction
Acronym: EROSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof. Dr., Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-2/8
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Sex Behavior; Ovarian Failure
Keywords: Ovarian Reserve; Sexual Satisfaction
MeSH Terms: conditions — Sexual Behavior; Orgasm | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Survey Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Other): All patients will be enrolled in one arm
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Patients will fill a questionary with 8 questions.

SUMMARY:
This is a survey study. The primary aim of the study is to investigate the relationship between the ovarian reserve and sexual satisfaction. All the patients who underwent ovarian reserve assessment for any reason will fill a questionnaire about sexual satisfaction. And the survey results will be compared with patients' ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to the gynecology clinic for any reason
* Patients with ovarian reserve tests
* 18-45 years

Exclusion Criteria:

* Mental disorders
* Anatomic genital malformations
* Patient' Decline to fill the survey
* Presence of malignancy
* Without any sexual activity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Sexual Satisfaction Score | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag University ART Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulahci Aslan E, Aslan K, Gurluler J, Uyaniklar O, Kilik T, Turk P, Ozden O, Kasapoglu I, Uncu G. EROSS study: effect of ovarian reserve on sexual satisfaction. J Obstet Gynaecol. 2022 Oct;42(7):3055-3060. doi: 10.1080/01443615.2022.2081798. Epub 2022 Jun 6. PMID 35666951